CLINICAL TRIAL: NCT06509945
Title: Allogeneic Peripheral Blood Stem Cell Transplantation as the First-line Treatment for Patients With the High-risk Peripheral T Cell Lymphoma
Brief Title: Allo-PBSCT as the First-line Treatment for Patients With the High-risk PTCL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-202404-PTCL
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: peripheral T cell lymphoma; allogeneic peripheral blood stem cell transplantation; high-risk
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention arm (Experimental): Participants will receive allogeneic peripheral blood stem cell transplantation.
  Interventions: Other: allogeneic peripheral blood stem cell transplantation

INTERVENTIONS:
Other: allogeneic peripheral blood stem cell transplantation — Patients achieved response to treatment will receive allogeneic peripheral blood stem cell transplantation.

SUMMARY:
This study is a single-center, single-arm, prospective phase II clinical trial that evaluates the efficacy and safety of allogeneic peripheral blood stem cell transplantation in the treatment of high-risk peripheral T-cells lymphoma patients achieved complete response (CR) or partial response (PR). Conventional conditioning regimen is adopted while the reduced-intensity conditioning regimens will be preferred. Donor hematopoietic stem cell infusion is performed on day 0. All patients will undergo bone marrow examination on day 14 and day 28 post-transplant, followed by bone marrow examinations every 30 days within the first year after transplantation, and every 60 days within the second year after transplantation. Positron emission tomography with 2-deoxy-2-[fluorine-18]fluoro-D-glucose integrated with computed tomography (18F-FDG PET/CT) imaging will be performed every 6 months after transplantation. If disease relapse is suspected during the follow-up period, bone marrow and relapse site examinations will be conducted at any time. The primary study endpoints are the 1-year and 2-year progression-free survival (PFS) rates post-transplant. Secondary study endpoints include the incidence of acute graft-versus-host disease (GVHD) within 180 days post-transplant, cumulative relapse rates at 1 year and 2 years post-transplant, 1-year and 2-year overall survival (OS), graft-versus-host disease-free, relapse-free survival (GRFS), non-relapse mortality (NRM), cumulative incidence of chronic GVHD, and the incidence of Cytomegalovirus （CMV）and Epstein-Barr virus（EBV）reactivation within 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and less than 70 years, regardless of gender 2. Peripheral T-cell lymphoma (PTCL) was diagnosed according to the 2016 WHO criteria and met any of the following criteria:

1. High risk: IPI（International Prognostic Index） score ≥ 3 or aaIPI（age-adjusted International Prognostic Index） score ≥ 2 ( aaIPI is suitable for patients younger than 60 years old).
2. Patients who achieved complete response (CR) or partial response (PR) after first-line chemotherapy (PET-CT or CT examination was performed according to the patient 's economic conditions） 3.Patients must have a suitable hematopoietic stem cell donor:

Related donors must have at least 5/10 matches for HLA-A, -B, -C, -DQB1, and - DRB1.

Unrelated donors must have at least 8/10 matches for HLA-A, -B, -C, -DQB1, and -DRB1.

4.Hematopoietic cell transplantation comorbidity index (HCT-CI) score ≤ 2. 5.ECOG (Eastern Cooperative Oncology Group) performance status: 0-2. 6.Adequate liver, kidney, and cardiopulmonary function, meeting the following requirements:

1. Serum creatinine ≤ 1.5x ULN (the upper limit of normal).
2. Cardiac function: Ejection fraction ≥ 50%.
3. Baseline oxygen saturation > 92%.
4. Total bilirubin ≤ 2.0 x ULN; ALT and AST ≤ 2.0 x ULN，AKP ≤ 2.0 x ULN
5. Pulmonary function: DLCO (corrected for hemoglobin) ≥ 40% and FEV1 (Forced Expiratory Volume in 1 second) ≥ 50%.

   7.Patients must have the ability to understand and be willing to participate in this study and sign an informed consent form.

   Exclusion Criteria:
   1. PTCL patients did not meet the criteria of high-risk.
   2. PTCL ALK + patients with CR after first-line treatment.
   3. History of malignancies other than lymphoid tumors within the 5 years prior to screening, except for adequately treated in situ cervical cancer, basal cell carcinoma, squamous cell carcinoma of the skin, and curatively treated localized prostate cancer or ductal carcinoma in situ
   4. ECOG ≥ 3.
   5. HCT-CI score ≥ 3.
   6. Any unstable systemic diseases, including but not limited to unstable angina, recent cerebrovascular accidents or transient ischemic attacks within the 3 months prior to screening, myocardial infarction within the 3 months prior to screening, congestive heart failure (New York Heart Association [NYHA] class ≥ III), severe arrhythmias requiring drug treatment after pacemaker implantation, significant liver, kidney, or metabolic diseases, and pulmonary arterial hypertension.
   7. Active, uncontrolled infections, including those associated with hemodynamic instability, new or worsening infection symptoms or signs, new infectious lesions on imaging, or persistent unexplained fever without signs or symptoms of infection.
   8. HIV-infected individuals.
   9. Active hepatitis B (HBV) or active hepatitis C (HCV) requiring antiviral therapy.
   10. History of autoimmune diseases
   11. Pregnant or breastfeeding women.
   12. Fertile males and females unwilling to use contraception during the treatment period and for 12 months after treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
1y and 2y-progression-free survival (PFS) | up to 1 years for the 1y-PFS and up to 2 years for the 2y-PFS
  1-year and 2-year progression-free survival (PFS) rates post-transplant

SECONDARY OUTCOMES:
acute graft-versus-host disease (aGVHD) | up to 180 days
  acute graft-versus-host disease (aGVHD) within 180 days post-transplant
1y and 2y-cumulative relapse rates (CIR) | up to 1 years for the 1y-CIR and up to 2 years for the 2y-CIR
  cumulative relapse rates (CIR) at 1 year and 2 years post-transplant
1y and 2y-overall survival (OS) | up to 1 years for the 1y-OS and up to 2 years for the 2y-OS
  overall survival (OS) at 1 year and 2 years post-transplant
graft-versus-host disease-free and relapse-free survival (GRFS) | up to 2 years
  graft-versus-host disease-free and relapse-free survival (GRFS) at 2 years post-transplant
non-relapse mortality (NRM) | up to 2 years
  non-relapse mortality (NRM) at 2 years post-transplant
cumulative incidence of chronic graft-versus-host disease (cGVHD) | up to 2 years
  cumulative incidence of chronic graft-versus-host disease (cGVHD) at 2 years post-transplant
Cytomegalovirus (CMV) and Epstein-Barr virus (EBV) reactivation | up to 1 year
  the incidence of CMV and EBV reactivation within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: xianmin Song, MD, Principal Investigator — Shanghai General HospitalShanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao C, Feng J, Gu H, Tang H, Xu L, Dong H, Dong B, Shu M, Bai Q, Liang R, Zhang T, Yang L, Wang Z, Chen X, Gao G. Distribution of lymphoid neoplasms in Northwest China: Analysis of 3244 cases according to WHO classification in a single institution. Ann Diagn Pathol. 2018 Jun;34:60-65. doi: 10.1016/j.anndiagpath.2017.05.005. Epub 2017 May 12. PMID 29661730
- [Background] Yang QP, Zhang WY, Yu JB, Zhao S, Xu H, Wang WY, Bi CF, Zuo Z, Wang XQ, Huang J, Dai L, Liu WP. Subtype distribution of lymphomas in Southwest China: analysis of 6,382 cases using WHO classification in a single institution. Diagn Pathol. 2011 Aug 22;6:77. doi: 10.1186/1746-1596-6-77. PMID 21854649